CLINICAL TRIAL: NCT01211210
Title: A Phase II/III Randomized Controlled Study of Neoadjuvant FOLFOX6 Treatment With or Without Radiation Compared to 5-Fu Based Chemoradiation in Treating Patients With Resectable Rectal Cancer
Brief Title: Neoadjuvant FOLFOX6 Chemotherapy With or Without Radiation in Rectal Cancer
Acronym: FOWARC
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanhong Deng, Doctor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GIHSYSU01
Record Dates: First submitted 2010-09-28; First posted 2010-09-29 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2013-11

CONDITIONS: Rectal Cancer
Keywords: rectal cancer; neoadjuvant therapy; oxaliplatin; radiation
MeSH Terms: conditions — Rectal Neoplasms | interventions — Fluorouracil; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A: 5Fu with Radiation (Active Comparator): Patients receive fluorouracil IV continuously and undergo radiotherapy once daily 5 days a week for 5-6 weeks.
  Interventions: Drug: fluorouracil
- B: FOLFOX with radiation (Experimental): Patients receive FOLFOX for 5 cycles and undergo radiotherapy as in arm I from the second cycle of FOLFOX
  Interventions: Drug: fluorouracil, oxaliplatin
- C: FOLFOX alone (Experimental): Patients receive FOLFOX for 4 cycles
  Interventions: Drug: fluorouracil, oxaliplatin

INTERVENTIONS:
Drug: fluorouracil — Drug: fluorouracil Given IV continuously Radiation: radiation therapy Given 5 days a week for 5-6 weeks
  Other Names: 5-Fu; RT
  Arms: A: 5Fu with Radiation
Drug: fluorouracil, oxaliplatin — Drug: fluorouracil Given IV continuously Drug: oxaliplatin Given IV Radiation: radiation therapy Given 5 days a week for 5-6 weeks
  Other Names: 5-Fu; Oxaliplatin; RT
  Arms: B: FOLFOX with radiation
Drug: fluorouracil, oxaliplatin — Drug: fluorouracil Given IV continuously Drug: oxaliplatin Given IV
  Other Names: 5-Fu; Oxaliplatin
  Arms: C: FOLFOX alone

SUMMARY:
RATIONALE: Preoperative 5-Fu based chemoradiation has become standard treatment for stage 2/3 rectal cancer. However whether these patients, especially T3N0-1M0 patients, really need radiation for local control after total mesentery excision being applied in routine practice is still unknown. And whether new drugs adding in can achieve better local and distant control is worth investigating.

PURPOSE: This randomized phase II trial is studying 5Fu based radiation therapy or FOLFOX based radiation or FOLFOX alone, comparing them to see how well they work when given before surgery in treating patients with intermediate risk resectable rectal cancer. It is not yet known whether 5-Fu based or FOLFOX based radiation therapy or even FOLFOX alone is more effective in treating rectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary Compare the objective response rate and the rate of local-regional relapse in patients with resectable rectal cancer treated with either 5-Fu or FOLFOX based chemoradiotherapy or FOLFOX alone without radiation.

Secondary

1. Compare the rate of pathologic complete response in patients treated with these regimens.
2. Compare the local recurrence rate

2.Determine the increase in the number of patients who are able to undergo sphincter-saving surgery after treatment with these regimens.

3.Correlate genetic patterns and the presence or absence of specific tissue biomarkers with response and prognosis in patients treated with these regimens.

4.Compare preoperative quality of life (QOL) of patients treated with oral capecitabine versus continuous infusion with fluorouracil. pelvic auto-nerve function 5.Determine the impact of oxaliplatin on neurotoxicity in patients treated with these regimens.

6.Compare the toxic effects of these regimens in these patients. 7.Compare the convenience of care in patients treated with these regimens. 8.Determine the impact of the type of surgical management on QOL at 1 year postoperatively in these patients.

OUTLINE: This is a randomized, multi-center study. Patients are stratified according to participating center, gender, clinical tumor stage (stage II vs. stage III), and surgical intent (sphincter saving vs. non-sphincter saving). Patients are randomized to 1 of 4 treatment arms.

* Arm A: Patients receive fluorouracil IV continuously and undergo radiotherapy once daily 5 days a week for 5-6 weeks.
* Arm B: Patients receive FOLFOX for 4 cycles and undergo radiotherapy as in arm I from the second cycle of FOLFOX.
* Arm C: Patients receive FOLFOX for 4 cycles Within 4-6 weeks after the completion of chemo radiotherapy, patients with responding or stable disease undergo surgery. Patients with progressive disease are treated at the discretion of the investigator and continue to be followed. Patients with progressive disease in arm III should received radiation.

Quality of life is assessed at baseline, at completion of chemo radiotherapy, and at 1 year after surgery.

After completion of study treatment, patients are followed every 3 months for 2 years, and then every 6 months for 3years.

PROJECTED ACCRUAL: A total of 495 patients will be accrued for this study within 5 years.

Eligibility Ages Eligible for Study: 18-75 Years old Genders Eligible for Study: Both Accepts Healthy Volunteers: No

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of adenocarcinoma of the rectum
2. Age: 18-75 years old
3. Stage of the primary tumor may be determined by ultrasound or MRI
4. Stage II (T_3-4, N_0 [N_0 is defined as all imaged lymph nodes < 1.0 cm]) OR stage III (T_1-4, N_1-2 [with the definition of a clinically positive lymph node being any node ≥ 1.0 cm]
5. Tumor palpable by digital rectal exam OR accessible by proctoscope or sigmoidoscope
6. Distal border of the tumor must be located < 12 cm from the anal verge
7. Tumor amenable to curative resection
8. 15 days prior recruit, meet the following criteria: Hematopoietic

   * Absolute neutrophil count ≥ 1,200/mm^3
   * Platelet count ≥ 100,000/mm^3 Hepatic
   * Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
   * Alkaline phosphatase ≤ 2 times ULN
   * AST ≤ 2 times ULN*
   * No hepatic disease that would preclude study treatment or follow-up
   * No uncontrolled coagulopathy Renal
   * Creatinine clearance > 50 mL/min
   * No renal disease that would preclude study treatment or follow-up
9. ECOG status: 0～1

Exclusion Criteria:

1. Hypersensitivity to fluorouracil, or oxaliplatin
2. No More than 4 weeks since prior participation in any investigational drug study
3. More than 4 weeks since prior participation in any investigational drug study
4. Clear indication of involvement of the pelvic side walls by imaging
5. With distant metastasis
6. History of invasive rectal malignancy, regardless of disease-free interval
7. Fertile patients must use effective contraception
8. Uncontrolled hypertension
9. Cardiovascular disease that would preclude study treatment or follow-up
10. Lack of upper gastrointestinal tract integrity or malabsorption syndrome，active upper gastrointestinal tract bleeding
11. Synchronous colon cancer
12. Pregnant or nursing, Fertile patients do not use effective contraception
13. Other malignancy within the past 5 years except effectively treated squamous cell or basal cell skin cancer, melanoma in situ, carcinoma in situ of the cervix, or carcinoma in situ of the colon or rectum
14. No psychiatric or addictive disorders, or other conditions that, in the opinion of the investigator, would preclude study participation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 495 (Actual)
Dates: Start 2010-06; Primary Completion 2017-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
3-year disease free survival | 2 years
  Compare 3-year disease free survival in patients with resectable rectal cancer treated with either 5-Fu or FOLFOX based chemoradiotherapy or FOLFOX alone without radiation.

SECONDARY OUTCOMES:
pathologic complete response rate | 1 years
local recurrence rate | 3 years
overall survival | 5 years
sphincter-saving surgery rate | 1 year
R0 resection rate | 1 year
predictive biomarkers | 3 year
quality of life | 3 year

CONTACTS AND LOCATIONS:
Overall Officials: Jianping Wang, MD, Study Director — Sun Yatsen University
Locations (1):
- Gastrointestinal Hospital, Sun Yatsen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Zhang T, Shi L, Jian L, Jiang J, Qiu Y, Xie F, Zhang J, Peng H, Zhong L, Chen Y, Zhong Y, Deng Y; FOWARC Group. Clinical Benefit and Cost-Effectiveness of FOLFOX Versus LCCRT in Neoadjuvant Treatment for Patients with Locally Advanced Rectal Cancer: An Economic Analysis of the FOWARC and PROSPECT Trial. Ann Surg Oncol. 2025 Dec 11. doi: 10.1245/s10434-025-18802-8. Online ahead of print. PMID 41379261
- [Derived] Wan H, Weng J, Cai J, Chen Z, Li P, Han J, Li Z, Wan Z, Yuan Z, Gan Y, Huang M, Li X, Li T, Liu X, Wang X, Yu H, Liu B, Lin J, Luo Y. Nodal Downstaging in Patients With Rectal Cancer: Survival Is Promising if YpN0 Is Achieved. Dis Colon Rectum. 2025 Oct 1;68(10):1162-1171. doi: 10.1097/DCR.0000000000003846. Epub 2025 Jul 8. PMID 40626521
- [Derived] Shi L, Zhang J, Deng Y. Associations of pretreatment emotional distress with adherence to therapy for patients with locally advanced rectal cancer: a post hoc analysis of the Chinese FOWARC phase 3 randomized clinical trial. BMC Med. 2025 May 21;23(1):293. doi: 10.1186/s12916-025-04128-5. PMID 40399932
- [Derived] Zhang J, Chi P, Shi L, Cui L, Gao J, Li W, Wei H, Cheng L, Huang Z, Cai G, Zhao R, Huang Z, Zhou H, Wei Y, Zhang H, Zheng J, Huang Y, Cai Y, Zhou Z, Kang L, Huang M, Wu X, Peng J, Ren D, Lan P, Wang J, Deng Y. Neoadjuvant Modified Infusional Fluorouracil, Leucovorin, and Oxaliplatin With or Without Radiation Versus Fluorouracil Plus Radiation for Locally Advanced Rectal Cancer: Updated Results of the FOWARC Study After a Median Follow-Up of 10 Years. J Clin Oncol. 2025 Feb 20;43(6):633-640. doi: 10.1200/JCO-24-01676. Epub 2024 Dec 13. PMID 39671537
- [Derived] Li L, Xu B, Zhuang Z, Li J, Hu Y, Yang H, Wang X, Lin J, Zhou R, Chen W, Ran D, Huang M, Wang D, Luo Y, Yu H. Accurate tumor segmentation and treatment outcome prediction with DeepTOP. Radiother Oncol. 2023 Jun;183:109550. doi: 10.1016/j.radonc.2023.109550. Epub 2023 Feb 21. PMID 36813177
- [Derived] Xie Y, Lin J, Wang X, Wang P, Zhuang Z, Zou Q, Cai D, Huang Z, Bai L, Tang G, Huang M, Wang J, Yu H, Luo Y. The Addition of Preoperative Radiation Is Insufficient for Lateral Pelvic Control in a Subgroup of Patients With Low Locally Advanced Rectal Cancer: A Post Hoc Study of a Randomized Controlled Trial. Dis Colon Rectum. 2021 Nov 1;64(11):1321-1330. doi: 10.1097/DCR.0000000000001935. PMID 33990500
- [Derived] Deng Y, Chi P, Lan P, Wang L, Chen W, Cui L, Chen D, Cao J, Wei H, Peng X, Huang Z, Cai G, Zhao R, Huang Z, Xu L, Zhou H, Wei Y, Zhang H, Zheng J, Huang Y, Zhou Z, Cai Y, Kang L, Huang M, Wu X, Peng J, Ren D, Wang J. Neoadjuvant Modified FOLFOX6 With or Without Radiation Versus Fluorouracil Plus Radiation for Locally Advanced Rectal Cancer: Final Results of the Chinese FOWARC Trial. J Clin Oncol. 2019 Dec 1;37(34):3223-3233. doi: 10.1200/JCO.18.02309. Epub 2019 Sep 26. PMID 31557064
- [Derived] Hu H, Huang J, Lan P, Wang L, Huang M, Wang J, Deng Y. CEA clearance pattern as a predictor of tumor response to neoadjuvant treatment in rectal cancer: a post-hoc analysis of FOWARC trial. BMC Cancer. 2018 Nov 20;18(1):1145. doi: 10.1186/s12885-018-4997-y. PMID 30458734
- [Derived] Qin Q, Ma T, Deng Y, Zheng J, Zhou Z, Wang H, Wang L, Wang J. Impact of Preoperative Radiotherapy on Anastomotic Leakage and Stenosis After Rectal Cancer Resection: Post Hoc Analysis of a Randomized Controlled Trial. Dis Colon Rectum. 2016 Oct;59(10):934-42. doi: 10.1097/DCR.0000000000000665. PMID 27602924
- [Derived] Deng Y, Chi P, Lan P, Wang L, Chen W, Cui L, Chen D, Cao J, Wei H, Peng X, Huang Z, Cai G, Zhao R, Huang Z, Xu L, Zhou H, Wei Y, Zhang H, Zheng J, Huang Y, Zhou Z, Cai Y, Kang L, Huang M, Peng J, Ren D, Wang J. Modified FOLFOX6 With or Without Radiation Versus Fluorouracil and Leucovorin With Radiation in Neoadjuvant Treatment of Locally Advanced Rectal Cancer: Initial Results of the Chinese FOWARC Multicenter, Open-Label, Randomized Three-Arm Phase III Trial. J Clin Oncol. 2016 Sep 20;34(27):3300-7. doi: 10.1200/JCO.2016.66.6198. Epub 2016 Aug 1. PMID 27480145
- [Derived] Huang M, Lin J, Yu X, Chen S, Kang L, Deng Y, Zheng J, Luo Y, Wang L, Lan P, Wang J. Erectile and urinary function in men with rectal cancer treated by neoadjuvant chemoradiotherapy and neoadjuvant chemotherapy alone: a randomized trial report. Int J Colorectal Dis. 2016 Jul;31(7):1349-57. doi: 10.1007/s00384-016-2605-7. Epub 2016 Jun 6. PMID 27270480